CLINICAL TRIAL: NCT02811380
Title: Evaluation of Safety and Performance of the BIP Central Venous Catheter With Anti-infective Coating
Brief Title: BIP CVC Clinical Safety and Performance Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bactiguard AB (Industry)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2535-2030-CDOC
Record Dates: First submitted 2014-12-23; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Surgery; Central Line Associated Blood Stream Infections (CLABSI)
Keywords: CVC; Healthcare associated infections (HAI); CLABSI; Noble metal alloy coating; CVC related thrombosis
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIP CVC (Experimental): Bactiguard Infection Protection Central Venous Catheter
  Interventions: Device: BIP CVC
- Uncoated standard CVC (Placebo Comparator): Uncoated standard Central Venous Catheter
  Interventions: Device: Uncoated Standard CVC

INTERVENTIONS:
Device: BIP CVC — BIP CVC catheterization to minimize risk of infections for venous access during and after elective large surgery
  Other Names: BIP Central Venous Catheter; Bactiguard coated CVC; Noble metal alloy coated Central Venous Catheter
  Arms: BIP CVC
Device: Uncoated Standard CVC — Standard CVC catheterization for venous access during and after elective large surgery
  Other Names: Standard CVC; Standard Central Venous Catheter; Uncoated CVC; Uncoated Central Venous Catheter
  Arms: Uncoated standard CVC

SUMMARY:
The primary objective of this trial was to determine Bactiguard coated BIP CVC's safety and performance and compare it to corresponding standard uncoated CVC.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the safety for the medical device of 'BIP central venous catheter". Safety is assessed by evaluation of adverse events (according to ISO 14155:2011). Examples of CVC related common events are phlebitis, infection at the infection site, catheter related bacteremia/fungemia, septicemia, sepsis, thrombosis, lung emboli and pneumothorax.

The secondary objective is to assess the overall performance by evaluating if there were any CVC handling problems experienced by the physician/health care personnel.

Furthermore, an exploratory objective of this study is to assess coating and microbial colonization.

Included in the study were men and women aged 18 years or older undergoing elective standardized large surgery with a planned CVC catheterization in right or left jugular vein or subclavian vein planned for at least 3 days.

This study is a single-centre, randomized, single-blind, controlled study of tolerability and safety of BIP CVC with noble metal alloy coating.

All statistical analyses is performed using the SAS® System, version 9.3 or higher (SAS Institute Inc., Cary, NC, USA). Data is to be summarized using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women ≥ 18 years of age
* Were, in the opinion of the investigator, able to communicate with and understand the trial personnel and comply with the requirements of the trial
* Requiring CVC catheterization for venous access, via right (most often) or left jugular vein or subclavian vein, during and after elective large surgery (liver or pancreas resection or intestinal/bowel surgery) planned for at least 3 days
* Had signed the informed consent

Exclusion Criteria:

* Known transmissive blood disease
* Known multiresistant bacterial colonization
* Ongoing infection
* Thromboembolism
* Anti-coagulation treatment excluding prophylaxis
* CVC during last 2 months
* History of problems with CVC
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Assessment of safety by evaluation of CVC related adverse events and any problems in post operative course. | Through study completion, an average of 10 days
  Overall assessment of safety by evaluation of CVC related adverse events and any problems in post operative course.

SECONDARY OUTCOMES:
Assessment of the overall performance | Through study completion, an average of 10 days
  Overall assessment of device performance by evaluation of any CVC handling problems experienced by the physician/health care personnel.

CONTACTS AND LOCATIONS:
Overall Officials: Sigridur Kalman, MD PhD Prof, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Dept. of Anesthesia and Intensive Care, Sweden, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No